CLINICAL TRIAL: NCT02669134
Title: CRT Improved Clinical Response UK Trial: A Multi-centre, Prospective, Randomized, Cross-over, Double Blind Study
Brief Title: CRT Improved Clinical Response UK Trial
Acronym: CRICKET
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: no record of study starting
Sponsor: Aston University (Other)
Collaborators: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 147-2015-PL
Record Dates: First submitted 2015-12-17; First posted 2016-01-29 (Estimated); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Cardiac Failure
Keywords: cardiac resynchronization therapy; optimization; heart failure; reverse left ventricular remodeling
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SonR optimization (Active Comparator): SonRtip bipolar atrial lead and LivaNova (Sorin) CRT-D implantation with device programming: SonR CRT Optimization programmed "AV+VV"
  Interventions: Other: Device programming
- Fixed settings (Placebo Comparator): SonRtip bipolar atrial lead and LivaNova (Sorin) CRT-D implantation with device programming device programming: sensed AV delay of 125 ms, VV delay of 0 ms (simultaneous); SonR CRT Optimization programmed "Off").
  Interventions: Other: Device programming

INTERVENTIONS:
Other: Device programming — SonRtip bipolar atrial lead and LivaNova (Sorin) CRT-D implantation with device programming: SonR CRT Optimization programmed "AV+VV"

SUMMARY:
The main objective of the CRICKET study is demonstrate that AV and VV optimization using SonR improves LV reverse remodeling response to CRT, compared with 'Fixed Settings' (FS) after 6 months of treatment. In this investigator-initiated, multi-centre, 2:2 factorial design, randomized, two-arm, double-blinded, cross-over, prospective trial, CRT recipients will be randomized to 'SonR' atrioventricular (AV) and ventricular-ventricular (VV) optimization or 'fixed settings'. The primary endpoint is an absolute reduction in left ventricular end-systolic volume.

DETAILED DESCRIPTION:
This is an investigator-initiated, multi-centre, 2:2 factorial design, randomized, two-arm, double-blinded, cross-over, prospective trial

Main study objectives

The main objective of the CRICKET study is demonstrate that AV and VV optimization using SonR improves LV reverse remodeling response to CRT, compared with 'Fixed Settings' (FS) after 6 months of treatment.

Study endpoints

Primary endpoint: The primary endpoint is a reduction (absolute difference) in LVESV with SonR vs FS after 6 months of treatment. The difference intra-patient of absolute change of LVESV value will be compared between two treatments: "SonR optimization" vs. "FS", defined as a sensed AV delay of 125 ms, VV delay of 0 ms (simultaneous).

Secondary endpoints:

Change in 6 MWT distance Change in NYHA class Change in quality of life Change in patient global assessment (EQ-5D) Change in Quality of life (MLWHF questionnaire) Change in LVEF AF burden Adverse Events

Number of subjects

Two hundred (200) patients will be enrolled. All patients will be implanted with the SonRtip bipolar atrial lead and a LivaNova (Sorin) CRT-D device offering both SonR optimization algorithm and atrio-biventricular pacing. Patients will be assigned to either the treatment or control arms, employing a 1:1 randomization with up to 100 patients in each of the 2 groups: Study Group (SonR CRT Optimization programmed "AV+VV") and Control Group ("Fixed Settings" (FS), defined as a sensed AV delay of 125 ms, VV delay of 0 ms (simultaneous); SonR CRT Optimization programmed "Off"). After the first 6 months, patients will be crossed-over to the alternative arm for another 6 months. There will be no washout period.

Duration of the clinical investigation

The study inclusion phase is expected to last approximately 1.5 years.

Follow-ups

Patients will be evaluated at baseline and randomized prior to implantation to SonR optimization or FS. A further clinical assessment, ECG and echocardiography will be undertaken at 6 months. At this point, patients will be crossed over to the other arm for another 6 months. The study closes following a further clinical and echocardiographic assessment at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for implantation of a CRT-D device according to current NICE or ESC guidelines;
* In sinus rhythm;
* NYHA class II, III or IV
* Have reviewed, signed and dated an informed consent

Exclusion Criteria:

* Inability to do a 6 min walk test.
* Previous implant with a pacemaker, an ICD or a CRT device (except upgrade from single chamber ICD with a fully functional defibrillation lead) not under recall or surveillance);
* Persistent atrial arrhythmias (or cardioversion for atrial fibrillation) within the past month;
* Ventricular tachyarrhythmia of transient or reversible causes such as acute myocardial infarction (MI), digitalis intoxication, drowning, electrocution, electrolyte imbalance, hypoxia or sepsis, uncorrected at the time of the enrolment;
* Incessant ventricular tachyarrhythmia;
* Unstable angina, or acute MI, Coronary Artery Bypass-Grafting (CABG), or Percutaneous Coronary Intervention (PCI) within the past 4 weeks;
* Correctable valvular disease that is the primary cause of heart failure;
* Indication for valve repair or replacement;
* Recent Cerebro-Vascular Accident (CVA) or Transient Ischemic Attack (TIA) (within the previous 3 months);
* On transplant waiting list;
* Previous heart transplant;
* Already included in another clinical study that could confound the results of this study;
* Life expectancy less than 1 year;
* Inability to understand the purpose of the study;
* Unavailability for scheduled follow-up or refusal to cooperate;
* Age of less than 18 years;
* Pregnancy;
* Drug addiction or abuse;
* Under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Left ventricular end-systolic volume (LVSV) | 6 months
  Reduction in LVESV with SonR vs FS after 6 months of treatment

SECONDARY OUTCOMES:
Walking distance on 6 -minute walk test | 6 months
  Change in 6 MWT distance
NYHA class | 6 months
  Change in NYHA class
Quality of life - general (non-disease specific) | 6 months
  Change in quality of life, assessed using EQ-5D (section 1)
Patient global assessment | 6 months
  Change in patient global assessment (included in EQ-5D, section 2)
Disease-specific quality of life (heart failure) | 6 months
  Change in quality of life (MLWHF questionnaire)
Left ventricular ejection fraction | 6 months
  Change in LVEF
AF burden | 6 months
  AF burden according to mode-switches
System safety assessed by Adverse Events | 6 months
  Report all Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Nichola Seare, PhD, Study Director — Aston University